CLINICAL TRIAL: NCT03044925
Title: Remote Magnetic Navigation-guided Ablation Versus Cryoablation for Persistent Atrial Fibrillation: A Prospective, Controlled Study
Brief Title: Remote Magnetic Navigation-guided Ablation Versus Cryoablation for Persistent Atrial Fibrillation (RECREATION Study)
Acronym: RECREATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qi Jin, Clinical Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20161404
Record Dates: First submitted 2017-01-30; First posted 2017-02-07 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; remote magnetic navigation; cryoablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cryosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote magnetic navigation (Experimental): Persistent atrial fibrillation ablation with remote magnetic navigation
  Interventions: Procedure: Remote magnetic navigation
- Cryoablation (Active Comparator): Persistent atrial fibrillation ablation with cryoballoon
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Remote magnetic navigation — Pulmonary vein isolation and other areas ablation guided by remote magnetic navigation
  Arms: Remote magnetic navigation
Procedure: Cryoablation — Pulmonary vein isolation and other areas ablation used by cryoballoon
  Arms: Cryoablation

SUMMARY:
Compare the safety and efficacy of remote magnetic navigation-guided ablation and cryoablation for patients with persistent atrial fibrillation.

DETAILED DESCRIPTION:
1. Compare the efficacy of remote magnetic navigation-guided ablation and cryoablation for patients with persistent atrial fibrillation.
2. Compare the safety of remote magnetic navigation-guided ablation and cryoablation for patients with persistent atrial fibrillation.
3. Compare the procedural parameters of remote magnetic navigation-guided ablation and cryoablation for patients with persistent atrial fibrillation.
4. Compare the effects of amiodarone on recurrence after these two different ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent atrial fibrillation (>7d, < 5years)
2. Age 18-75 years
3. Patient is mentally and linguistically able to understand the aim of the trial and to show sufficient compliance in following the trial protocol

Exclusion Criteria:

1. Any previous left atrial ablation or surgery
2. Any cardiac surgery or percutaneous coronary intervention within 3 months prior to enrollment
3. Stroke or transient ischemic attack within 6 months prior to enrollment
4. Myocardial infarction within 3 months prior to enrollment
5. Anteroposterior left atrial diameter > 55 mm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy (time to first AF recurrence after blanking period) | one year
  the time to first AF recurrence after blanking period (month)
Clinical safety (Any procedure-related complications) | one year
  Any procedure-related complications

SECONDARY OUTCOMES:
Procedure time (min) | one week
Time to first cardiovascular hospitalization (month) | one year
QoL of 12 months (Units on a Scale) | one year
X-ray time (min) | one week

CONTACTS AND LOCATIONS:
Overall Officials: Qi Jin, MD, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Result] Kuck KH, Furnkranz A, Chun KR, Metzner A, Ouyang F, Schluter M, Elvan A, Lim HW, Kueffer FJ, Arentz T, Albenque JP, Tondo C, Kuhne M, Sticherling C, Brugada J; FIRE AND ICE Investigators. Cryoballoon or radiofrequency ablation for symptomatic paroxysmal atrial fibrillation: reintervention, rehospitalization, and quality-of-life outcomes in the FIRE AND ICE trial. Eur Heart J. 2016 Oct 7;37(38):2858-2865. doi: 10.1093/eurheartj/ehw285. Epub 2016 Jul 5. PMID 27381589
- [Result] Kuniss M, Greiss H, Pajitnev D, Akkaya E, Deubner N, Hain A, Bodammer L, Berkowitsch A, Chierchia GB, Hamm CW, Neumann T. Cryoballoon ablation of persistent atrial fibrillation: feasibility and safety of left atrial roof ablation with generation of conduction block in addition to antral pulmonary vein isolation. Europace. 2017 Jul 1;19(7):1109-1115. doi: 10.1093/europace/euw146. PMID 27738068
- [Result] Jin QI, Pehrson S, Jacobsen PK, Chen XU. Efficacy and Safety of Atrial Fibrillation Ablation Using Remote Magnetic Navigation: Experience from 1,006 Procedures. J Cardiovasc Electrophysiol. 2016 Mar;27 Suppl 1:S23-8. doi: 10.1111/jce.12929. PMID 26969219